CLINICAL TRIAL: NCT07057492
Title: A Prospective Multicenter Clinical Study on the Long-term Prognosis of Patients With ST-segment Elevation Myocardial Infarction Using Cardiac Magnetic Resonance Imaging.
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); Beijing Chao Yang Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); First People's Hospital of Yulin (Other); Wuhan Asia Heart Hospital (Other); Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Qian geng, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: 2018QG-CMR
Record Dates: First submitted 2025-07-02; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2018-01

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST-segment elevation Myocardial Infarction；cardiac magnetic resonance; prediction model
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the development cohort: The development cohort consisted of STEMI patients from four major medical centers, all of whom received primary PCI treatment and underwent cardiac magnetic resonance imaging. This cohort served as the basis for constructing the prognostic prediction model.
- the external validation cohort: The external validation cohort comprised STEMI patients from four additional medical centers, all of whom underwent primary PCI and subsequent cardiac magnetic resonance imaging. This independent cohort was used to evaluate the model's generalizability and predictive performance in diverse clinical settings.

SUMMARY:
This prospective, multicenter study was designed to develop and validate a risk prediction model for major adverse cardiovascular events (MACE) in patients with acute ST-segment elevation myocardial infarction (STEMI) based on cardiac magnetic resonance (CMR) parameters.

From January 2018 to December 2023, consecutive acute STEMI patients who underwent primary percutaneous coronary intervention (PCI) were enrolled across eight participating medical centers. Baseline clinical characteristics were systematically collected, and all patients underwent CMR examination 5-7 days after PCI to assess myocardial injury and functional parameters. The primary composite endpoint, MACE, included cardiovascular death, recurrent myocardial infarction, hospitalization for heart failure, and unplanned revascularization.

To ensure robust model development and validation, the study assigned patients from four centers to form the development cohort, while those from the other four centers constituted the external validation cohort. Predictive variables were initially screened using least absolute shrinkage and selection operator (LASSO) regression, followed by multivariable Cox proportional hazards regression to identify independent predictors. A nomogram was subsequently constructed to provide individualized risk stratification. Model performance was evaluated in terms of discrimination (C-index, ROC analysis), calibration (calibration curves), and clinical utility (decision curve analysis).

This study aims to develop a CMR-based prediction model to better identify high-risk STEMI patients, providing clinicians with valuable tools for early intervention and personalized management.

ELIGIBILITY:
Inclusion Criteria: Patients were required to meet the diagnostic criteria for STEMI, defined as elevated serum cardiac biomarkers (troponin) above the 99th percentile upper reference limit, accompanied by at least one of the following: 1.Chest pain lasting >30 minutes; 2.ST-segment elevation ≥0.1 mV in two or more contiguous limb leads or ≥0.2 mV in two or more contiguous precordial leads on 12-lead electrocardiography. Additional inclusion criteria: Age >18 years; First-time STEMI treated with primary PCI; Management strategy compliant with current clinical guidelines; Killip class ≤III; Willingness to undergo CMR examination and clinical follow-up.

Exclusion Criteria:Patients were excluded if they had contraindications to CMR, including implanted cardiac pacemakers, claustrophobia, gadolinium contrast allergy, or renal insufficiency. Additional exclusions comprised those with Killip class IV heart failure or clinically unstable conditions, as well as concomitant valvular disease, congenital heart disease, pulmonary hypertension, or persistent atrial fibrillation-conditions known to confound cardiac structural/functional assessments. We also excluded individuals with prior myocardial infarction, PCI, or coronary artery bypass grafting (CABG) to ensure a first-event STEMI cohort. Finally, patients with psychiatric/neurocognitive disorders impairing compliance, or those with poor-quality or incomplete CMR sequences, were not enrolled.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary PCI-treated patients with acute STEMI
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | From enrollment through the 3-year follow-up completion
Major Adverse Cardiovascular Events | From enrollment to the 3-year follow-up completion

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China